CLINICAL TRIAL: NCT03747536
Title: Ipratropium Bromide Spray as Treatment for Sialorrhea in Children: a Randomized, Double-blind, Placebo-controlled Crossover Study
Brief Title: Ipratropium Bromide Spray as Treatment for Sialorrhea in Children
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Peng You, Principle Investigator, Department of Otolaryngology Head and Neck Surgery, Western University, London Health Sciences Centre
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LondonHSC
Record Dates: First submitted 2018-11-14; First posted 2018-11-20 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Sialorrhea
Keywords: Ipratropium bromide; Sialorrhea; Pediatric
MeSH Terms: conditions — Sialorrhea | interventions — Ipratropium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study drug will be dispensed as a metered-dose spray bottle of ipratropium bromide or identical placebo prepared by the Hospital Pharmacy. Clinician, investigator, care provider, as well as outcome assessor will be blinded to the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): ipratropium bromide administered via metered dose spray (21 micrograms per spray). 1-2 spray sublingual or to buccal mucosa every 6 hours up to 4 times a day
  Interventions: Drug: Ipratropium bromide
- Placebo (Placebo Comparator): normal saline administered via metered dose spray. 1-2 spray sublingual or to buccal mucosa every 6 hours up to 4 times a day
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ipratropium bromide — ipratropium bromide via metered dose spray (21 micrograms per spray)
  Other Names: Atrovent
  Arms: Intervention
Other: Placebo — normal saline delivered via metered dose spray
  Arms: Placebo

SUMMARY:
Double-blind, clinical trial investigating the effects of ipratropium spray versus placebo spray in children with sialorrhea

DETAILED DESCRIPTION:
Excess drooling, or sialorrhea, is a chronic problem seen in pediatric patients with oral-motor dysfunction or neurodevelopmental abnormalities. Despite significant social and physical detriment from sialorrhea, an effective and safe treatment remains elusive.

The investigator's objective is to study the effect of sublingual ipratropium (an anticholinergic aerosol spray) on sialorrhea in the pediatric population

Method: A double-blind, randomized, placebo-controlled cross-over trial of sublingual ipratropium bromide application in pediatric patients with inappropriate drooling. Patients are recruited from the sialorrhea clinic and informed consent is obtained. Patients are randomized to receive ipratropium bromide, 1- 2 metered doses (sprays) of active drug (21 micrograms per metered dose) or matching placebo, every 6 hours up to a maximum of 4 times per day, in a double-blind, cross-over design using randomization tables. Total treatment length is two weeks for each limb of the study with a 2 week washout period. The primary outcome measure is the reporting of sialorrhea using a validated scales. Secondary outcome includes global assessment of treatment, patient satisfaction, and adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents aged 5-18 with a history of excessive drooling

Exclusion Criteria:

* known hypersensitivity to ipratropium bromide
* surgery for sialorrhea within one year
* the concurrent use of acetylcholinesterase inhibitors, cholinergic agents, or anticholinergic agents
* botulinum toxin for drooling within the preceding six months
* a history of glaucoma
* the presence of clinically significant urinary retention or outflow obstruction as evidenced by patient history or documented urodynamic studies

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-10-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Drooling Severity and Frequency Scale | Change from baseline sialorrhea at 2 weeks following each treatment arm
  Also referred to as the Thomas Stonell and Greenberg scale. This is a validated tool using patient reported scores for drooling severity and frequency. Drooling severity is scored on a scale with minimum value of 1 and maximum value of 5. A higher value represents a worse outcome. The frequency is scored on a scale with minimum value of 1 and maximum value of 4. A higher value represents a worse outcome. The subscales (severity and frequency) can be interpreted independently or combined through addition to compute a total score.
Change in Drooling impact scale | Change from baseline sialorrhea at 2 weeks following each treatment arm
  The drooling impact scale is a validated self-administered questionnaire used to measure saliva-control in children. The scale consists of 10 questions/subscales, each with a minimum score of 1 and a maximum score of 10. For all subscales, the higher value represents a worse outcome. The total score is reported and is calculated by adding the score of all 10 subscales.

SECONDARY OUTCOMES:
Patient Global Impression of Improvement Scale | At start of trial and weekly self recording up to 8 weeks
  The Patient Global Impression of improvement scale is a single 7-point scale that requires the patient/caregiver to assess how much the illness has improved or worsened relative to a baseline state at the beginning of the intervention. The minimum score is 1 and the maximum score is 7. A higher value represents a worse outcome. To be collected through patient booklet
Adverse effect | Intermittent up to 8 weeks
  Documentation of all adverse effects encountered during study period
Patient feedback | Weekly self recording up to 8 weeks.
  Open ended patient comment related to the intervention. To be collected through patient booklet

CONTACTS AND LOCATIONS:
Overall Officials: Julie Strychowsky, MD, Principal Investigator — London Health Science Centre

IPD SHARING:
Plan to Share IPD: Undecided